CLINICAL TRIAL: NCT06045832
Title: MAXPOWER Biological Antibacterial Liquid Oral Helicobacter Pylori Eradication Evaluation
Brief Title: Oral Helicobacter Pylori Eradication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-017
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: H. Pylori Infection
Keywords: Oral H. pylori; Eradication Evaluation; Antibiotic-free; Mouthwash
MeSH Terms: interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: At the beginning of the study, the demographic characteristics of the study participants were recorded in detail, including sex, age, history of smoking, alcohol consumption, presence of bad breath and GI symptoms. After that, a randomization list was generated using SPSS (version 25.0), and the included patients were randomized in a 1:1 ratio according to the randomization table to receive either MAXPOWER Biological Antibacterial Liquid gargle treatment (Gargle 3 times a day for 2 min each time for 7 days) or gargle with water (Gargle 3 times a day for 2 min each time for 7 days). Then, all patients were retested for oral H. pylori.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): At the beginning of the study, the demographic characteristics of the study participants are recorded in detail, including sex, age, history of smoking, alcohol consumption, presence of bad breath and GI symptoms. The patients who are randomized into control group receive water gargle treatment (Gargle 3 times a day for 2 min each time for 7 days) Then, all patients were retested for oral H. pylori using H. pylori saliva test.
  Interventions: Device: Water
- MAXPOWER Biological Antibacterial Liquid group (Active Comparator): At the beginning of the study, the demographic characteristics of the study participants are recorded in detail, including sex, age, history of smoking, alcohol consumption, presence of bad breath and GI symptoms. The patients who are randomized into MAXPOWER Biological Antibacterial Liquid group receive MAXPOWER Biological Antibacterial Liquid gargle treatment (Gargle 3 times a day for 2 min each time for 7 days) Then, all patients were retested for oral H. pylori using H. pylori saliva test.
  Interventions: Device: MAXPOWER Biological Antibacterial Liquid

INTERVENTIONS:
Device: MAXPOWER Biological Antibacterial Liquid — MAXPOWER Biological Antibacterial Liquid is a mouthwash product self-developed in China, which contains betaine, antibacterial peptide and other antimicrobial substances, which have been proved by experiments to have a good biological safety and at the same time have a killing effect on bacteria. Mouthwash belongs to the category of medical devices, not drugs.
  Arms: MAXPOWER Biological Antibacterial Liquid group
Device: Water — Water
  Arms: Control group

SUMMARY:
Helicobacter pylori (H. pylori) is a serious health threat that infects approximately half of the global population. In addition to colonizing the stomach, H. pylori has been shown to survive in the oral microenvironment and is associated with a variety of oral diseases, gastric eradication failure, and reinfection. Currently, traditional systemic antibiotic therapy has little effect on oral H. pylori, and mouthwashes available on the market for oral H. pylori eradication often contain multiple antibiotics or complex essential ingredients, which can cause unpredictable effects on the human body. Therefore, there is an urgent need for a mouthwash that does not contain antibiotics and is effective against oral H. pylori. This study focuses on the eradication effect of MAXPOWER Biological Antibacterial mouthwash on oral H. pylori in a population.

DETAILED DESCRIPTION:
Inclusion criteria: oral H. pylori-positive patients, verified by H. pylori saliva test (HPS),aged 18-70 years visiting the outpatient clinic of Changhai Hospital from March 1, 2023, to August 1, 2023, were enrolled.

Exclusion criteria: (1) Zollinger-Ellison syndrome, gastric cancer, upper gastrointestinal bleeding, or active peptic ulcer; (2) the coexistence of significant concomitant illnesses, including heart diseases, renal failure, hepatic disease, previous abdominal surgery, lactation or pregnancy; and (3) not willing to participate in the study.

Written informed consent was obtained from all patients prior to participation in the study.

ELIGIBILITY:
Inclusion Criteria:Oral H. pylori-positive patients, verified by H. pylori saliva test (HPS),aged 18-70 years visiting the outpatient clinic of Changhai Hospital from March 1, 2023, to August 1, 2023, were enrolled.

Exclusion Criteria: (1) Zollinger-Ellison syndrome, gastric cancer, upper gastrointestinal bleeding, or active peptic ulcer; (2) the coexistence of significant concomitant illnesses, including heart diseases, renal failure, hepatic disease, previous abdominal surgery, lactation or pregnancy; and (3) not willing to participate in the study.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Oral H. pylori eradication rate | 7 days
  We tested patients for oral H. pylori using H. pylori saliva test (HPS) to .HPS is a lateral flow immunochromatographic test device that uses saliva as testing sample detecting oral H. pylori within few minutes. The principle of HPS is based on monoclonal antibody react with oral urease produced by H. pylori.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Contact us to obtain the IPD

REFERENCES:
- [Background] Yee JKC. Are the view of Helicobacter pylori colonized in the oral cavity an illusion? Exp Mol Med. 2017 Nov 24;49(11):e397. doi: 10.1038/emm.2017.225. PMID 29170474
- [Derived] Lai Y, Dong X, Song Y, Zhao J, Du Y, Li Z. Novel MAXPOWER biological antibacterial liquid for eradicating oral Helicobacter pylori. BMC Infect Dis. 2024 May 29;24(1):540. doi: 10.1186/s12879-024-09424-8. PMID 38811871